CLINICAL TRIAL: NCT05752565
Title: Physical Activity and FVIII Elimination: Relevance to Personalized Therapy in Severe Hemophilia A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, De Cristofaro Raimondo, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2364
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- patients with severe HA under FVIII concentrates prophylaxis (Other): patients with severe HA under FVIII concentrates prophylaxis
  Interventions: Device: SenseWear armband device

INTERVENTIONS:
Device: SenseWear armband device — Device: SenseWear armband device Metabolic Holter, Physical Activity and Lifestyle, Portable outpatient "multi-sensor" energy consumption in calories (EE), movement, physical activity, quality of life

SUMMARY:
In persons with severe haemophilia A infused factor VIII half-life and other pharmacokinetic can vary according to determinants such as blood group, von Willebrand factor (VWF) level or age. However, FVIII pharmacokinetics (PK) has not been throughly studied in patients with severe HA as a function of daily physical activity. It si known that vigorous intensity physical activity/exercise can transiently but significantly increase circulating levels of endogenous VWF and consequently FVIII in normal subjects and in patients with moderate or mild haemophilia A. The proposed study is a Proof of Concept one as it will be aimed at investigating the relation between daily physical activity, measured by Sensewear armband device, as number of daily steps and PK variability of infused rec-FVIII concentrate. This kind of investigation has never been done and it is a great interest also for the evaluation of patient's qualitiy of life.

DETAILED DESCRIPTION:
In persons with severe haemophilia A infused factor VIII half-life and other pharmacokinetic can vary according to determinants such as blood group, von Willebrand factor (VWF) level or age. However, FVIII pharmacokinetics (PK) has not been throughly studied in patients with severe HA as a function of daily physical activity. It si known that vigorous intensity physical activity/exercise can transiently but significantly increase circulating levels of endogenous VWF and consequently FVIII in normal subjects and in patients with moderate or mild haemophilia A. The proposed study is a Proof of Concept one as it will be aimed at investigating the relation between daily physical activity, measured by Sensewear armband device, as number of daily steps and PK variability of infused rec-FVIII concentrate. This kind of investigation has never been done and it is a great interest also for the evaluation of patient's qualitiy of life. Physical Examinations at screening and subsequent study visits a physical examination will be performed on the following body systems being described as normal or abnormal: general appearance, headand neck, eyes and ears, nose and throat, heart, abdomen, extremities and joints, lymph nodes and neurological. At screening, if an abnormal condition is detected, the condition will be described on the medical history CRF. At study visit, if a new abnormal or worsened abnormal pre-existing condition is detected, the condition will be described n the CRF.

ELIGIBILITY:
Inclusion Criteria:

* patients 12-60 yo with severe HA under FVIII concentrates prophylaxis will be selected at the Haemostasis and Thrombosis Center of the Fondazione Policlinico Gemelli IRCCS Rome (FPG)

Exclusion Criteria:

* all patients with malignant tumors or
* patietnts treated with anticoagulant / antiplatelet agents
* patients suffering from other congenital coagulation disorders (von Willebrand disease, other congenital deficiency of coagulation factors or severe thrombocytopenia (< 30,000 Plt/uL)

Ages: 12 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Study of the association between physical activity, measured by mean nuber of daily steps, with the Area Under the Curve (AUC) PK parameter in patients with severe HA under prophylaxis. | 12 months
  Study of the association between physical activity, measured by mean nuber of daily steps, with the Area Under the Curve (AUC) PK parameter in patients with severe HA under prophylaxis. Investigate whether and how the daily physical activity (measured as number of steps, using the SenseWear Armband device) affects the PK parameter. .
Association PK parameter and number of daily steps | 12 months
  In more details the study aims to evaluate whether and how the FVIII PK parameter is significantly associated with the mean number of daily steps in patients with severe HA

CONTACTS AND LOCATIONS:
Locations (1):
- FPG, Roma, Italy